CLINICAL TRIAL: NCT06576557
Title: Knowledge Translation and Exercise for Degenerative Meniscal Tears and Early Osteoarthritis: the KNEE-DEeP Feasibility Study
Brief Title: Knowledge Translation and Exercise for Degenerative Meniscal Tears and Early Osteoarthritis: KNEE-DEeP Study
Acronym: KNEE-DEeP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0000
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee; Meniscus; Degeneration
Keywords: Health Care Quality, Access, and Evaluation; Feasibility Studies; Exercise Therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KNEE-DEeP Intervention arm (Experimental): The KNEE-DEeP study delivers an intervention at both the level of the healthcare professional and the patient. Healthcare professionals (GPs and physiotherapists) will receive a educational workshop and resources to use with patient participants. Patients in the intervention arm will receive an 'enhanced consultation' with their GP and early access to a 'best practice' one-hour physiotherapy session in University Hospital Kerry, along with educational resources.
  Interventions: Other: KNEE-DEeP intervention- Knowledge translation and exercise for early degenerative knee pain

INTERVENTIONS:
Other: KNEE-DEeP intervention- Knowledge translation and exercise for early degenerative knee pain — The intervention for health care professionals (GPs and physiotherapists) will consist of training and education. The two-hour educational workshop for GPs will focus on diagnosis and management of patients with early degenerative knee pain, and enhancing communication skills. Training for physiotherapists will focus on delivery of a 'best practice' session. The patient participant intervention will consist of an 'enhanced consultation' delivered by the GP. This will involve a physical exam, key educational messages, written information and a treatment plan. Patients will receive a single session of physiotherapy within 2 weeks of referral from their GP. This 'best practice' session will focus on self-management skills, targeted patient education, goal setting, action planning and exercise prescription.

SUMMARY:
Knee pain due to a degenerative meniscal tear (DMT) or early osteoarthritis (OA) is a frequent presentation in middle-aged and older adults. In the knee joint a DMT can occur normally with age, but is also associated with the continuum of knee OA. Exercise is recommended as the main treatment to aid recovery, while an arthroscopy (camera in the knee) to remove torn cartilage does not provide any additional benefit. Despite this many patients in Ireland with this type of knee pain are referred to an orthopaedic surgeon by their GP, and do not receive recommended care from their physiotherapist.

The first phase of this project designed the KNEE-DEeP (Knowledge Translation and Exercise for Early Degenerative Knee Pain) intervention to deliver better care to patients with DMT and early OA. The overall aim of this feasibility study is to test the KNEE-DEeP intervention to ensure it can be delivered as planned and it is acceptable to patients, and health care professionals (HCPs) involved in intervention delivery; GPs and physiotherapists. This is in preparation for carrying out a larger future trial.

As part of the intervention, GPs and physiotherapists will receive an educational workshop. Patient participants in turn will receive an 'enhanced consultation' from their participating GP and a 'best practice' physiotherapy session focusing on strategies to enhance self-management. This approach will be tested out by enrolling 15 GPs, five physiotherapist and 36 patients in the feasibility study. Patients will be followed up after 12 weeks and six months to track their progress. As part of the evaluation all GPs, physiotherapists and patients will complete questionnaires and a sub-set will provide more in-depth feedback via interviews conducted over the phone or online.

DETAILED DESCRIPTION:
KNEE-DEeP Intervention Design

The KNEE-DEeP intervention was designed to address modifiable barriers at the patient, provider and system level to evidence based care for DMT and early OA. According to the Medical Research Council's guidance on the development and evaluation of complex healthcare interventions a multi-component strategy is needed to address these barriers, using the best available evidence and appropriate theory.

The intervention was designed using the Behavioural Change Wheel (BCW) eight-step process. The Theoretical Domains Framework (TDF) was used to identify relevant determinants of change and develop an in-depth understanding of each target behaviour. The KNEE-DEeP intervention will target both GPs and physiotherapists, and their patients with early OA and DMT. GPs will receive a training workshop and educational resources to facilitate an enhanced clinical consultation about this type of knee pain. Given the emphasis placed by Irish GPs on timely access to physiotherapy in managing this condition, early access to a single 'best practice' session of physiotherapy will be a key component of the patient intervention to address this service-level barrier. The content of the patient intervention delivered by the GP and physiotherapist will be underpinned by clinical practice guidelines, stakeholder input and the evidence base on management of chronic knee pain.

Specific KNEE-DEeP study objectives are:

1. Determine the acceptability of the intervention content and delivery to HCPs and patients
2. Determine adherence of GPs and physiotherapists to study processes around intervention delivery to patients
3. Assess fidelity related to intervention delivery and intervention receipt, from the perspectives of HCPs and patients.
4. Determine if data collection procedures and outcome measures are feasible and acceptable to HCPs and patients
5. Determine feasibility of HCP and patients' recruitment and retention procedures
6. Investigate the magnitude of change and variability in the clinical outcome measures

Study Design and Setting

The KNEE-DEeP study is a non-randomised feasibility study that includes an embedded mixed methods process evaluation. Assessments will be performed at baseline, 12 weeks (primary endpoint) and 24 weeks. Recruitment is anticipated to last 6 months, with each patient participant taking part in the trial for 6 months and the last follow-up due 12 months after the start of recruitment.

Set in general practices in Kerry and North Cork and in the Physiotherapy Department of University Hospital Kerry (UHK), a publicly funded hospital also in the South-West of Ireland.

A single arm feasibility study was chosen rather than a comparative design because the main focus was to resolve uncertainties about the acceptability and feasibility of the intervention itself, and its mode of delivery. A non-randomised design was deemed suitable as it was an opportunity to test the intervention with a greater number of HCP and patient participants.

Sample Size

As this is a feasibility study, a formal sample size calculation has not been carried out.

ELIGIBILITY:
Inclusion Criteria for Participants with Knee Pain:

* Attended their GP with an episode of non-traumatic knee pain
* Have knee pain attributed to a DMT or early degenerative changes based on the GP's clinical assessment (this standardised assessment is a component of the GP training)
* Aged between 35 and 69 years inclusive

Exclusion Criteria:

* Recent trauma likely to be associated with considerable tissue damage
* Fulfilling the American College of Rheumatology clinical classification criteria for knee OA (these criteria reflect later signs of OA or established disease)
* Moderate or advanced knee OA on x-ray (or Kellgren-Lawrence x-ray score ≥ Grade 3)
* Having an acutely swollen or locked knee, or suspected ligament injury on physical exam
* Inflammatory arthritis
* Surgery or significant trauma of the index knee within the previous 2 years
* Pregnancy
* Unable to communicate in English
* Preference for accessing physiotherapy treatment privately prior to the 'best practice' session.

Inclusion Criteria for Participating GPs (n=15) and Physiotherapists (n=5):

* Eligible GPs will be working in practices within traveling distance (< 50 km) of University Hospital Kerry and willing to attend a two-hour training workshop
* Eligible physiotherapists will be involved in the delivery of outpatient musculoskeletal physiotherapy services at University Hospital Kerry and available to participate in training to deliver the 'best practice' physiotherapy intervention

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in physical function from baseline to 12 weeks as measured by Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS) | Baseline and 12 weeks
  This 7-item measure of physical function is derived from the activities of daily living and sport/recreation subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS). Psychometric testing shows the KOOS-PS to be valid and reliable for use in groups with knee OA, making it an suitable tool for measuring knee-related function in this research. Scores range from 0 (extreme problems) to 100 (no problems).

SECONDARY OUTCOMES:
Change in physical function from baseline to 12 weeks as measured by Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS) | Baseline and 24 weeks
  This 7-item measure of physical function is derived from the activities of daily living and sport/recreation subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS). Psychometric testing shows the KOOS-PS to be valid and reliable for use in groups with knee OA, making it an suitable tool for measuring knee-related function in this research. Scores range from 0 (extreme problems) to 100 (no problems).
Change in knee pain from baseline to 12 weeks as measured by Knee Injury and Osteoarthritis Outcome Score Pain Subscale | Baseline and 12 weeks
  This nine item subscale of the KOOS is scored (0 to 100) and reported individually. The KOOS subscales are valid, responsive and reliable questionnaires and has been used extensively knee OA and knee arthroscopy trials.
Change in knee pain from baseline to 24 weeks as measured by Knee Injury and Osteoarthritis Outcome Score Pain Subscale | Baseline and 24 weeks
  This nine item subscale of the KOOS is scored (0 to 100) and reported individually. The KOOS subscales are valid, responsive and reliable questionnaires and has been used extensively knee OA and knee arthroscopy trials.
Change in pain self-efficacy from baseline to 12 weeks as measured by the Pain Self-efficacy (PSEQ 2-item short form) | Baseline and 12 weeks
  The 2 items identified from the PSEQ reflect confidence in one's ability to work and lead a normal life despite pain and are scored on a 7-point Likert scale from "Not at all confident" (0) to "Completely confident" (6), with scores ranging from 0 to 12 to perform activity despite pain. This 2-item shortened form of the PSEQ is a valid, responsive and reliable questionnaires and has been used extensively in chronic musculoskeletal disorders research.
Change in pain self-efficacy from baseline to 24 weeks as measured by the Pain Self-efficacy (PSEQ 2-item short form) | Baseline and 24 weeks
  The 2 items identified from the PSEQ reflect confidence in one's ability to work and lead a normal life despite pain and are scored on a 7-point Likert scale from "Not at all confident" (0) to "Completely confident" (6), with scores ranging from 0 to 12 (maximal confidence) to perform activity despite pain. This 2-item shortened form of the PSEQ is a valid, responsive and reliable questionnaires and has been used extensively in chronic musculoskeletal disorders research.
Change in fear avoidance beliefs from baseline to 12 weeks as measured by the physical activity subscale of the Fear Avoidance Belief Questionnaire (FABQ) | Baseline and 12 weeks
  This four-item physical activity sub-scale of the FABQ quantifies the level of fear about physical activity. While primarily studied in patients with low-back pain, it is a reliable scale to measure fear avoidance beliefs in knee OA.
Change in fear avoidance beliefs from baseline to 24 weeks as measured by the physical activity subscale of the Fear Avoidance Belief Questionnaire (FABQ) | Baseline and 24 weeks
  This four-item physical activity sub-scale of the FABQ quantifies the level of fear about physical activity. While primarily studied in patients with low-back pain, it is a reliable scale to measure fear avoidance beliefs in knee OA.
Change in health related quality of life from baseline to 12 weeks as measured by the EuroQol Five-Dimensional Questionnaire (EQ-5D-5L) | Baseline and 12 weeks
  Health-related quality of life will be measured with this generic health index, which comprises five dimensions of health (mobility, self-care, usual activities, pain or discomfort, anxiety or depression) and a Visual Analogue Scale (VAS) of current overall health status ranging from 0 (worst
  imaginable health) to 100 (best imaginable health).
Change in health related quality of life from baseline to 24 weeks as measured by the EuroQol Five-Dimensional Questionnaire (EQ-5D-5L) | Baseline and 24 weeks
  Health-related quality of life will be measured with this generic health index, which comprises five dimensions of health (mobility, self-care, usual activities, pain or discomfort, anxiety or depression) and a Visual Analogue Scale (VAS) of current overall health status of current overall health status ranging from 0 (worst
  imaginable health) to 100 (best imaginable health).
Patient Satisfaction with Care at 12 weeks | 12 weeks
  Participants will be asked to rate "overall satisfaction with the care you received in this study" using a 7-point scale ranging from "extremely unsatisfied" to "extremely satisfied"
Adherence to exercise and physical activity plan at 12 weeks | 12 weeks
  Adherence to the exercise and physical activity plan agreed with the physiotherapists will be rated by the patient participant via questionnaire scored on an 11-point Numerical Rating Scale (0 = not at all and 10 = completely as instructed).
Use of health care and co-interventions for knee pain from baseline to 12 weeks | 12 weeks
  A self-report checklist completed will record visits to health care providers (additional physiotherapy and GP consultations, other health professional or secondary care consultations), injection use, complementary therapies, use of prescription and over-the-counter medication, imaging, other participation in structured exercise between baseline and 12 weeks
Use of health care and co-interventions for knee pain from 12 to 24 weeks | 24 weeks
  A self-report checklist completed will record visits to health care providers (additional physiotherapy and GP consultations, other health professional or secondary care consultations), injection use, complementary therapies, and imaging between 12 and 24 weeks
Change in pain medication from baseline to 12 weeks | 12 weeks
  Change in pain medication use from baseline to 12 weeks will be assessed with a 7-point Likert scale (much less to much more).

OTHER OUTCOMES:
Feasibility of the intervention as rated by patient participants at 12 weeks using the Feasibility of Intervention Measure (FIM) | 12 weeks
  The FIM is a 4-item scale that measures the extent to which a new intervention can be successfully delivered within a given setting. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean.
Feasibility of the intervention with clinician (physiotherapist and GP) participants as measured using the Feasibility of Intervention Measure (FIM) | 12 weeks
  The FIM is a 4-item scale that measures the extent to which a new intervention can be successfully delivered within a given setting. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). A mean score is calculated.
The acceptability of the intervention to patient participants will be measured at 12 weeks using the Theoretical Framework of Acceptability (TFA) | 12 weeks
  Generic questionnaire adapted to assess KNEE-DEeP intervention acceptability from the perspectives of intervention recipients measured using a five-point Likert scale from 'Strongly disagree' to 'Strongly agree
The acceptability of the intervention to HCP (physiotherapist and GP) participants will be measured at 12 weeks using the Theoretical Framework of Acceptability (TFA) | 12 weeks
  Generic questionnaire adapted to assess KNEE-DEeP intervention acceptability from the perspectives of intervention recipients, measured using a five-point Likert scale from 'Strongly disagree' to 'Strongly agree
Fidelity of delivery and receipt of the KNEE-DEeP GP 'enhanced consultation' will be assessed by a checklist completed by the GP (fidelity of delivery) and patient (fidelity of receipt) at baseline (0 weeks) | Baseline
  Bespoke checklist documenting the key elements of the GP 'enhanced consultation'
Fidelity of delivery of the KNEE-DEeP physiotherapy 'best practice' session will be assessed by a bespoke checklist completed by the physiotherapist post-intervention delivery | Immediately post-intervention
  Bespoke checklist documenting the key elements of the physiotherapy 'best practice' session
Qualitative data on intervention acceptability and feasibility will be collected via semi-structured interviews with patient participants | No fixed timepoint, qualitative data will be collected between 2 weeks and 8 weeks post intervention receipt
  A twenty minute interview conducted online or via telephone question will explore participants experience of the intervention. A subset of patients will be invited to interview.
Qualitative data on intervention acceptability and feasibility will be collected via semi-structured interviews with a sub-set of participating health care professionals (GP and physiotherapists) | No fixed timepoint, qualitative data will be collected from health care professionals after at least 3-month of study participation
  A twenty minute interview conducted online or via telephone question will explore participants experience of the intervention, both receiving the educational workshop and training and delivering the patient intervention
Adverse events reported to the research team will be recorded in an adverse events log throughout the duration of the study | Duration of the study and followup period (approx 12 months)
  Adverse events can be reported to the research team by participating GPs, physiotherapists of patients. Defined as any problem that participants believe was caused by the intervention (exercise or advice) and required them to seek treatment and/or lasted for two or more days.

CONTACTS AND LOCATIONS:
Overall Officials: Helen O'Leary, BSc Physio, Principal Investigator — University of Limerick; Karen McCreesh, BSc Physio, Study Chair — University of Limerick
Locations (1):
- University Hospital Kerry, Tralee, Kerry, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request once the study has been completed. Available dataset will consist of anonymised IPD relating to patient clinical outcome measures. Due to the small number of participating clinicians, data gathered from participating clinicians will not be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 6 months after planned papers have been published (quantitive x 1 and qualitative x ). Data will remain available for 60 months
Access Criteria: All requests from qualified researchers engaging in independent scientific research will be considered, and will be provided following review and approval of a research proposal. Access can be requested by contacting the principal investigator helen.oleary@ul.ie

REFERENCES:
- [Background] Culvenor AG, Oiestad BE, Hart HF, Stefanik JJ, Guermazi A, Crossley KM. Prevalence of knee osteoarthritis features on magnetic resonance imaging in asymptomatic uninjured adults: a systematic review and meta-analysis. Br J Sports Med. 2019 Oct;53(20):1268-1278. doi: 10.1136/bjsports-2018-099257. Epub 2018 Jun 9. PMID 29886437
- [Background] Siemieniuk RAC, Harris IA, Agoritsas T, Poolman RW, Brignardello-Petersen R, Van de Velde S, Buchbinder R, Englund M, Lytvyn L, Quinlan C, Helsingen L, Knutsen G, Olsen NR, Macdonald H, Hailey L, Wilson HM, Lydiatt A, Kristiansen A. Arthroscopic surgery for degenerative knee arthritis and meniscal tears: a clinical practice guideline. BMJ. 2017 May 10;357:j1982. doi: 10.1136/bmj.j1982. No abstract available. PMID 28490431
- [Background] Bhattacharyya T, Gale D, Dewire P, Totterman S, Gale ME, McLaughlin S, Einhorn TA, Felson DT. The clinical importance of meniscal tears demonstrated by magnetic resonance imaging in osteoarthritis of the knee. J Bone Joint Surg Am. 2003 Jan;85(1):4-9. doi: 10.2106/00004623-200301000-00002. PMID 12533565
- [Background] Keavy R, Horton R, Al-Dadah O. The prevalence of musculoskeletal presentations in general practice: an epidemiological study. Fam Pract. 2023 Feb 9;40(1):68-74. doi: 10.1093/fampra/cmac055. PMID 35747902
- [Background] O'Leary H, Ryan LG, Robinson K, Conroy EJ, McCreesh K. "You'd be better off to do the keyhole and make a good job of it" a qualitative study of the beliefs and treatment expectations of patients attending secondary care with degenerative meniscal tears. Musculoskelet Sci Pract. 2021 Feb;51:102281. doi: 10.1016/j.msksp.2020.102281. Epub 2020 Oct 27. PMID 33161307
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Background] Wood G, Neilson J, Cottrell E, Hoole SP; Guideline Committee. Osteoarthritis in people over 16: diagnosis and management-updated summary of NICE guidance. BMJ. 2023 Jan 24;380:24. doi: 10.1136/bmj.p24. No abstract available. PMID 36693668
- [Background] Perruccio AV, Stefan Lohmander L, Canizares M, Tennant A, Hawker GA, Conaghan PG, Roos EM, Jordan JM, Maillefert JF, Dougados M, Davis AM. The development of a short measure of physical function for knee OA KOOS-Physical Function Shortform (KOOS-PS) - an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 May;16(5):542-50. doi: 10.1016/j.joca.2007.12.014. Epub 2008 Feb 21. PMID 18294869
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Nicholas MK, McGuire BE, Asghari A. A 2-item short form of the Pain Self-efficacy Questionnaire: development and psychometric evaluation of PSEQ-2. J Pain. 2015 Feb;16(2):153-63. doi: 10.1016/j.jpain.2014.11.002. Epub 2014 Nov 14. PMID 25463701
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Sekhon M, Cartwright M, Francis JJ. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC Health Serv Res. 2022 Mar 1;22(1):279. doi: 10.1186/s12913-022-07577-3. PMID 35232455
- [Background] Hurst NP, Kind P, Ruta D, Hunter M, Stubbings A. Measuring health-related quality of life in rheumatoid arthritis: validity, responsiveness and reliability of EuroQol (EQ-5D). Br J Rheumatol. 1997 May;36(5):551-9. doi: 10.1093/rheumatology/36.5.551. PMID 9189057
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] O'Leary H, Robinson K, Glynn L, Lenehan B, McCreesh K. "You're stuck in the middle here": a qualitative study of GPs' experiences of managing knee pain attributed to a degenerative meniscal tear. BMC Prim Care. 2023 Jun 21;24(1):127. doi: 10.1186/s12875-023-02075-9. PMID 37344762
- [Derived] O'Leary H, Toomey C, Ryan LG, Robinson K, Glynn L, French HP, McCreesh K. Knowledge translation and exercise for degenerative meniscal pathology and early osteoarthritis (KNEE-DEeP): Protocol for a single arm feasibility study. HRB Open Res. 2025 Jan 24;8:14. doi: 10.12688/hrbopenres.14049.1. eCollection 2025. PMID 40028467